CLINICAL TRIAL: NCT06440395
Title: Small Steps for Big Changes: Implementing an Evidence-Based Diabetes Prevention Program Into Diverse Urban Communities
Brief Title: Small Steps for Big Changes - Healthy Cities Implementation Science
Acronym: HCIS
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Public Health Agency of Canada (PHAC) (Other Government); McMaster University (Other); Memorial University of Newfoundland (Other); Brock University (Other); Arthritis Research Centre of Canada (Other)
Responsible Party: Principal Investigator, Mary Jung, Associate Professor, University of British Columbia
Other Study IDs: H23-01930
Record Dates: First submitted 2024-05-13; First posted 2024-06-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: PreDiabetes
Keywords: Implementation Science; Exercise Behaviour; Diet Behaviour; Adherence; Health Behaviour Change
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Small Steps for Big Changes: Diabetes Prevention Program: Diabetes Prevention Program (one-treatment group) The diabetes prevention program is a 4-week program that will introduce participants to a regular healthy behaviours that includes exercise and simple dietary strategies. There is no randomization to this program - all individuals enrolled will partake in the same program and will be followed up for 24 months after the program has concluded.
  Interventions: Behavioral: Behavioural: Small Steps for Big Changes Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Behavioural: Small Steps for Big Changes Diabetes Prevention Program — The 4-week behaviour change program will introduce participants to a regular healthy lifestyle including exercise and dietary changes for reducing sugar intake, reducing refined/processed carbohydrate intake, increasing vegetable consumption. The 4-week program will include six supervised exercise sessions and three exercise sessions performed independently (e.g., at home or outside of the YMCA). The supervised session will include brief behavioural counselling sessions that teach participants self-regulatory skills to promote independence and long-term adherence to exercising and dietary changes.

SUMMARY:
Small Steps for Big Changes (SSBC) is a diet and exercise counselling program that significantly reduces the risk of developing Type 2 Diabetes (T2D). In partnership with YMCAs in Canada spanning 8 provinces, the aim of this study is to scale-up program delivery and evaluate the implementation and effectiveness of SSBC. To evaluate implementation, the number of staff trained/patients enrolled, attendance, sessions delivered as planned, delivery costs, and number of sites continuing to deliver the program will be examined. To evaluate program effectiveness, changes in patient health (e.g., T2D status, blood glucose, weight, exercise, diet) will be measured over 2 years following program completion.

DETAILED DESCRIPTION:
In partnership with YMCAs in Canada spanning 8 provinces (overseeing 44 distinct community facilities/sites), the investigators will adapt and deliver our evidence-based diabetes prevention program, Small Steps for Big Changes. The purpose of this project is to evaluate the implementation and effectiveness of SSBC across diverse urban communities.

Specifically, the investigators aim to:

1. Evaluate the implementation and sustainability of the program by examining the number of staff trained/patients enrolled, attendance, sessions delivered as planned, delivery costs, and number of sites continuing to deliver the program.
2. Examine clinical-effectiveness of the program on: T2D status (self-report and HbA1c; primary outcomes), cardiorespiratory fitness, anthropometric (weight, waist circumference, resting heart rate), health behaviours (exercise, diet).
3. Examine cost-effectiveness of the program on: healthcare resource utilization, and health-related quality of life (secondary outcomes).

Research Design:

A hybrid type 2 implementation-effectiveness study design (Curran et al., 2012) with multi/mixed methods will be used to evaluate the implementation and effectiveness of SSBC.

SSBC program:

SSBC will be administered and facilitated by the community facility trainers at YMCA locations. SSBC consists of 6 sessions delivered over 4 consecutive weeks, with each session comprising brief (20-30 mins) counselling that support participants self-regulatory skills to promote independence and long-term adherence to healthy dietary behaviours and regular exercise, followed by 20-30 mins of supervised aerobic exercise.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Community-dwelling adults aged 18 years or older
* able to read and speak English
* has prediabetes assessed by one of the following means: (a) physician-diagnosed prediabetes, (b) HbA1c values between 5.7 - 6.4% (American Diabetes Association, 2012), (c) an American Diabetes Association risk questionnaire score indicating increased risk (>5)
* Individuals who have previously been diagnosed with type 2 diabetes but who are in remission (defined as achieving glycated hemoglobin (A1C) of < 6.4% without any diabetes-related medications for a minimum of 3 months) will be eligible to participate.

Exclusion Criteria:

- Patients currently diagnosed type 2 diabetes with an HbA1c of 6.5% or greater.

Organizational partners

Inclusion criteria:

- Senior leadership and/or management of our Canadian YMCA delivery partner organizations

Exclusion criteria: N/A

Site leads/managers

Inclusion criteria:

- YMCA staff who manage/coordinate programs (e.g., general manager of health programs) for each site willing to act as SSBC site lead champion.

Exclusion criteria: N/A

Coaches

Inclusion criteria:

Site staff certified as SSBC coaches to deliver the program.

Exclusion criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators aim to recruit a community-based sample of adults at risk of type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 4400 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes status | 0, 12, and 24 months post intervention
  Self reported HbA1c%
Change in HbA1c | 0, 12 and 24 months post intervention
  Venipuncture blood collection of HbA1c% through laboratory testing in a subsample of participants
Adoption of SSBC | 0, 52, 104, 156, 208 weeks
  Proportion and representativeness of coaches and implementation support team obtained through program records
Reach of SSBC | 0, 52, 104, 156, 208 weeks
  Proportion of patients' enrolled and completing the intervention, proportion of implementation staff trained and retained. Demographics of the patients and staff
Dose Delivered | During delivery of the intervention
  Number of SSBC sessions delivered by coaches (0-6) will be gathered through coach checklists
Fidelity of SSBC delivery | During delivery of the intervention
  Frequency with which clients recieve each core component and quality of counselling skills measured using session checklists.
Number of adaptations of SSBC | Prior to, and throughout delivery of the intervention (0-104 weeks), sustainment planning and delivery (104-208 weeks)
  Number of adaptations made prior to delivery of SSBC and during SSBC delivery. Number of adaptations needed for sustainment and during sustainment. Adaptation information will be gathered through meeting minutes with site leads, annual reports from delivery sites and through interviews with coaches and site leads.
Types of adaptations of SSBC | Prior to, and throughout delivery of the intervention (0-104 weeks), sustainment planning and delivery (104-208 weeks)
  Type of adaptations made prior to delivery of SSBC and during SSBC delivery. Adaptation information will be gathered through meeting minutes with site leads, annual reports from delivery sites and through interviews with coaches and site leads.
Receptivity to SSBC among patients' and staff | 4, and 52 weeks (patients), during delivery (staff)
  Patient acceptability and satisfaction will be assessed using the 1-item net promoter score, overall satisfaction measure developed in house and the theoretical framework of acceptability measure. Interviews will be conducted with a subsample of patients at each site (2-3 per site) after completing SSBC. Staff satisfaction and burden will be assessed using brief surveys a various points through the program delivery with coaches (baseline, after 5, 10, 20 clients) and site leads (baseline and at the end of SSBC delivery). Satisfaction and acceptability will also be examined among staff using qualitative interviews.
Cost of Delivering SSBC | 104, 156, 208 weeks
  Costs incurred for implementing SSBC at the delivery sites will be collected through annual reporting from the delivery sites.
Membership rates | 104, 156, 208 weeks
  The proportion of individuals who convert their one-month free pass to a facility membership and the retention of this membership over time will be calculated. This information will be collected from annual reports from delivery sites and client surveys.

SECONDARY OUTCOMES:
Change in body weight | 0, 4, 52, and 104 weeks
  Measured in pounds
Change in cardiorespiratory fitness | 0, 4, 52, and 104 weeks
  Distance walked in the six minute walk test will be conducted at sites with access to a walking track.
Change in physical activity behaviour using the Godin Leisure Time Physical Activity Questionnaire | 0, 4, 52, and 104 weeks
  The Godin Leisure Time Physical Activity Questionnaire will be used to examine physical activity behaviour. Respondents report the frequency of strenuous, moderate, and mild physical activity for bouts of 15 or more minutes during a 7-day period. The scores are multiplied by weigths and summed into an overall score reports in metabolic equivalents of task (METs)/minutes of physical activity per week.
Changes in physical activity using the 2-item Physical Activity Vital Signs measure | 0, 4, 52, and 104 weeks
  The 2-item Physical Activity Vital Signs measure will be used to collect information on physical activity behaviour. Two questions are self-reported: 1) "How many days during the past week have you performed physical activity where your heart beats faster and your breathing is harder than normal for 30 minutes or more?" and 2) "How many days in a typical week do you perform activity such as this?" The responses are reported as days during the past week over days in a typical week, with scores ranging from 0 to 7 for each question.
Change in dietary intake | 0, 4, 52, and 104 weeks
  Assessed using the brief food frequency questionnaire. Participants are asked about their intake of five foods within the past week: fruits, vegetables, sweets, bread and rice/pasta. Items are rated on a 6-point scale. The questionnaire also uses a composite score for refined carbohydrates (sum of bread and rice/pasta).
Determinants of intervention implementation | 52 weeks
  Aspects of the larger social, political and economic environment that may influence delivery of the adapted intervention will be assessed by interview. These interviews will also gather qualitative data potential factors that impact delivery of SSBC at the site including context, acceptability, adaptability, feasibility, compatibility, cost, culture, complexity and self efficacy. These interviews will be conducted among coaches and managerial staff.
Sustainability outcomes and determinants | 104, 156 and 208 weeks
  Data will be collected on the number of sites continuing delivery, the number of coaches continuing delivery, the number of clients run through SSBC and the number of implementation strategies that are utilized. This data will be gathered through program records. Focus groups will be conducted at each site over the 2-year sustainability phase to gather information on the contextual factors that impact sustainment outcomes.
Change in health-related quality of life (EQ-5D-5L Profile) | 0, 4, 52, and 104 weeks
  The EQ-5D-5L consists of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Participants are asked to indicate their level of functioning (from 1 "no problems" to 5 "extreme problems") on each of the five dimensions of the EQ-5D-5L. The EQ-5D-5 L describes 3125 distinct health states, with 11111 representing the best and 55555 the worst possible health states. The Canadian EQ-5D-5 L scoring algorithm will be applied to generate index scores which range from - 0.148 for the worst (55555) to 0.949 for the best (11111) health states.
Change in health-related quality of life (EQ-5D-5L Visual Analogue Scale) | 0, 4, 52, and 104 weeks
  Health status will be assessed with the EQ-5D-5L visual analogue scale. Participants report on their health on a visual analogue scale from 0 (worst health) to 100 (best health)
Change in health resource utilization | 0, 52, and 104 weeks
  The extent to which participants use medical services will be assessed using the Health Resource Utilization Survey. The information will be combined with the EQ-5D-5L health related quality of life profiles to calculate the cost-effectiveness of the program.

OTHER OUTCOMES:
Organizational readiness | 0 weeks
  Organizational readiness for change measured by the Organizational Readiness for Implementing Change (Shea et al., 2014)
Change in 24-hour movement | 0, 4, 52, 104 weeks
  Change in 24-hour movement will be examined using a 4-item measure to collect information on time spent in activity, sitting and sleeping in hours and minutes
Change in waist circumference | 0, 4, 52, and 104 weeks
  Measured at level of Iliac crest in centimetres by the coach
Baseline self-compassion | 0 weeks
  Patients' self-compassion will be assessed at baseline using the short form self-compassion scale (Raes et al., 2011). This 12-item measure has participants rate the extent to which they engage in certain behaviours on a 5-point response scale from 1 (almost never) to 5 (almost always). Sub scales can be computed by adding item scores. A total self-compassion score is computed.

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (12):
  - Castle Downs Family YMCA, Edmonton, Alberta
  - Health and Exercise Psychology Laboratory, Kelowna, British Columbia
  - Prince George Family YMCA, Prince George, British Columbia
  - Tong Louie Family YMCA, Surrey, British Columbia
  - YMCA of Brandon Health and Fitness Centre, Brandon, Manitoba
  - Elmwood-Kildonan, Winnipeg, Manitoba
  - Saint John Regional Y, Saint John, New Brunswick
  - Ches Penney Family YMCA, St. John's, Newfoundland and Labrador
  - John W. Lindsay YMCA, Halifax, Nova Scotia
  - YMCA 3 Rivers, Kitchener, Ontario
  - YMCA of Greater Toronto - Scarborough Health and Fitness Centre, Scarborough Village, Ontario
  - YMCA of Regina Health, Fitness and Aquatics Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weatherson K, Bourne JE, Cranston K, Braaten K, Grieve N, Kelly J, Jung ME. Scaling Up a Diabetes Prevention Program in Geographically and Ethnoculturally Diverse Urban Regions of Canada: Protocol for a Hybrid Type 2 Implementation-Effectiveness Study. JMIR Res Protoc. 2026 Jan 19;15:e80276. doi: 10.2196/80276. PMID 41553750